CLINICAL TRIAL: NCT04264936
Title: A Open-label, Single-arm, Phase Ib/II Study of RC48-ADC and JS001 to Evaluate the Safety and Pharmacokinetics of Subjects With Locally Advanced or Metastatic Urothelial Cancer
Brief Title: A Study of RC48-ADC(Antibody Drug Conjugate) and JS001 to Evaluate the Safety and Pharmacokinetics of Subjects With Locally Advanced or Metastatic Urothelial Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C014
Record Dates: First submitted 2020-01-15; First posted 2020-02-11 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC and JS001 (Experimental)
  Interventions: Drug: RC48-ADC and JS001

INTERVENTIONS:
Drug: RC48-ADC and JS001 — Recombinant Humanized anti-HER2(Human epidermal growth factor receptor-2) Monoclonal Antibody-MMAE(Monomethyl Auristatin E) Conjugate For Injection and JS001 Injection

SUMMARY:
This is an open-label, single-arm, Phase Ib/II investigator-initiated trial of RC48-ADC combined with JS001 to evaluate the safety and pharmacokinetics of subjects with locally advanced or metastatic urothelial cancer

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form; Aged 18 years and above; ECOG(Eastern Cooperative Oncology Group) performance is 0 or 1; Life expectancy greater than 12 weeks; Patients with locally advanced or metastatic malignant urothelial carcinoma which is platinum naive and cisplatin ineligible, or progressed after at least one line standard systemic chemotherapy (including progression within 12 months of neo-/adjuvant therapy);

Cisplatinum ineligible patients should meet one of the following criteria:

1. Aged 70 years and above, and ECOG performance is 1;
2. Serum creatinine >= 1.0xULN or CrCl<60ml/min;
3. Lose of hearing >= Grade 2;
4. Peripheral nerve disorder >= Grade 2 Patients with measurable and appreciable tumor lesions according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1); Willing to provide primary lesion samples for the purpose of PD-L1 and HER2 tests.

Adequate organ function as defined by the following criteria:

1. absolute neutrophil count(ANC) >= 1.5 x 10^9/L;
2. platelets>=100* 10^9/L;
3. Total serum creatinine <=1.5*ULN;
4. serum aspartate transaminase (AST) and serum alanine transaminase (ALT) <=2.5*upper limit of normal (ULN), or AST and ALT<=5*ULN if liver function abnormalities are due to underlying malignancy; normal serum creatinine ;
5. Left ventricular ejection fraction (LVEF) >=50%
6. Hemoglobin>=9g/dl Women of child-bearing potential and men must agree to use adequate contraception (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete sexual abstinence, or sterilized partner) prior to study entry and during the period of therapy and for 30 days after the last dose of study drug;

Exclusion Criteria:

* Allergy to RC48-ADC, or JS001, or their components Received anti-cancer therapy including chemotherapy, radiotherapy, immunotherapy or other clinical trial treatments within 3 weeks of starting study treatment Unresolved toxicities from prior anti-cancer therapy, except for alopecia Previously treated with HER2-ADC and/or anti-PD-1 or anti-PD-L1 or anti PD-L2 therapies; Underwent major surgery within 4 weeks of first dose of study drug and not completely recovered; Received vaccine within 4 weeks of first dose of study drug Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or greater than or equal to Class 2 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study; History of other neoplastic disease within 3 years prior to the study drug, with exception of resolved/curable cancers such as basal skin cancer or squamous cell skin cancer,.

Metastasis to CNS(central nervous system) and/or carcinomatous meningitis, with exception for the patients who received treatment of metastasis to CNS and/or carcinomatous meningitis and had stable disease for at least 3 months, and no evidence of progression within 4 weeks of first dose of study treatment. No evidence of new or expanded metastasis, and untreated with radiotherapy, surgery or steroid therapy within 4 weeks of first dose of study treatment.

History of allogeneic hematopoietic stem cell transplantation or organ transplantation; Patients who had received systemic steroid therapy within the last 2 years; Pregnancy or lactation; Positive results of HIV testing; Active HBV(hepatitis B virus) or HCV(hepatitis C virus) infection Active tuberculosis; Other disorders with clinical significance according to the researcher's judgment; Unwilling or unable to participate in all required study evaluations and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | through study completion, an average of 1 year
  rate of adverse events
maximal tolerated dose | through study completion, an average of 1 year
  dose-limiting toxity

SECONDARY OUTCOMES:
Peak Plasma Concentration(Cmax) | through study completion, an average of 1 year
  Maximum observed plasma concentration
Immunogenicity | through study completion, an average of 1 year
  Numbers of participants with anti-drug antibody positive
objective response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first；assessed up to 60 months
  evaluated by RECIST 1.1 every 8 weeks
the area under the curve (AUC) | through study completion, an average of 1 year
  Area under the plasma concentration versus time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No